CLINICAL TRIAL: NCT07181733
Title: Exploring B-Type Natriuretic Peptide (BNP) Evolution, From the Neonatal to Adolescent Period, as a Tool to Early Identify the Risk for Metabolic Syndrome (MetS) in a Former Preterm and Full Term Adolescent Population
Brief Title: BNP in Pediatric Metabolic Syndrome
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Alessia Claudia Codazzi, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: BNP-MetS
Record Dates: First submitted 2025-03-03; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Syndrome
Keywords: adolescent; BNP
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- subjects adolescents, born preterm/IUGR
- subjects adolescents, born at term

SUMMARY:
MetS is a syndrome characterized by a combination of diabetes, hypertension and visceral obesity, altered blood lipids, beginning in childhood, leading to chronic disease in adulthood. Adult criteria for defining MetS require a minimum of 3 risk factors, listed in the NCEP ATP III (National Cholesterol Education Program, Adult Treatment Panel III, ATP III), they are hyperglycaemia, hypertriglyceridemia, low HDL-C, hypertension, obesity and increased waist circumference.

The pediatric definitions are described mainly by Cooks, Zimmet and de Ferranti are as well based on the presence of ≥ 3 symptoms: obesity (BMI) , waist circumference, glucose intolerance, dyslipidaemia (high triglycerides and/or low HDL-C), High BP. Pediatric criteria of MetS are not univocally defined and symptoms may be fluctuant in adolescent period, therefore the prevalence ranges from 4.2%13 to 9.2%. A number of researchers have used factor analysis of MetS components to develop a risk score to identify children at higher risk for developing MetS. Several MetS risk factors have origins during the prenatal and early postnatal period. In particular, it is known that preterm newborns are more prone to develop this condition once adults, but little is known about the adolescent transition, particularly, in Italy.

From 2008 - 2011, thirty-four full-term and 36 premature infants were studied, evaluating echocardiographic parameters and BNP concentrations during the first month of life. In this population, now adolescents, it was decided to measure BNP, both current and previous values, in order to verify whether this parameter can be associated with MetS and meet the need to identify high-risk children.

Adolescents affected by MetS were defined on the basis of the available literature: they must present ≥ 3 of the following signs: hyperglycaemia, dyslipidaemia (triglycerides and HDL-C), arterial hypertension, obesity (BMI and waist circumference). Other blood parameters were also evaluated as associated factors, such as white blood cell count, glycosylated haemoglobin, creatinine, urea nitrogen, and suPAR. Doppler echocardiography and tissue Doppler parameters, psychosocial variables (KIDSCREEN-10).

BNP has been shown to play a role not only in heart disease but also in adult patients with obesity, insulin resistance, and diabetes, all of which are present in MetS. Therefore, the primary objective is to assess whether BNP can be an index associated with adolescent MetS. The opportunity was taken to evaluate a population of premature and full-term adolescents. BNP was previously studied in the first month of life, and it is possible to establish a correlation with the adolescent situation. Therefore, the cohort of newborns who are now between 13 and 15 years of age will be recalled.

The data available in the literature and clinical experience suggest a prevalence of metabolic syndrome of between approximately 5 and 10%.

ELIGIBILITY:
Inclusion Criteria:

* adolescents whose BNP concentration and echocardiographic parameters analysed during their first month of life (2009-11)

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients whose BNP concentration and echocardiographic parameters was analysed during their first month of life (2009-11) of life at Fondazione IRCCS Policlinico San Matteo
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Association of BNP with MetS in adolescent period | December 2025
  we define MetS when an adolescent presents 3 of the following symptoms: hyperglycemia (>110 mg/dl), dyslipidemia (triglycerides <= 120 mg/dl and/or HDL-C < 60 mg/dl), High BP (systolic >120 mmHg diastolic >80 mmHg) , obesity (BMI > 30 and waist circumference > 0.5).

SECONDARY OUTCOMES:
association of BNP in neonatal period and adolescents biomedical measurements | December 2025
Association of adolescent BNP and MetS within categories of psychosocial variables (as identified by the KIDSCREEN-10 instrument) which are established to have a role in the development of MetS | December 2025
  Psychosocial data:
  KIDSCREEN-10 instrument: Self-report questionnaire for the assessment of adolescents' subjective health and health-related quality of life (HRQOL). The normalized score will be then categorized with a cut-off of 50.
Association of BNP in neonatal period with MetS | December 2025

CONTACTS AND LOCATIONS:
Locations (1):
- U.O.S. Cardiologia Pediatrica, Pavia, pavia, Italy

IPD SHARING:
Plan to Share IPD: No